CLINICAL TRIAL: NCT00572052
Title: Comparison of Glycemic Control Achieved With a 31 Gauge x 6 mm NovoFine® Needle vs. a BD 29 Gauge x 12.7 mm Ultra-Fine® Needle in Subjects With Diabetes Mellitus and a BMI Exceeding 30 kg/m2: An Open Label, Randomized, Two-Period Crossover Study
Brief Title: Comparison of Glycemic Control Achieved With 2 Different Needles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEEDLEN-2168
Record Dates: First submitted 2007-12-04; First posted 2007-12-12 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NovoFine® needle 6 mm
Device: Ultra-Fine needle 12.7 mm

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to investigate if a 31 gauge x 6 mm needle will provide comparable blood glucose control to the 29 gauge x 12.7 mm needle in obese subjects with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Current treatment with insulin or insulin analogues for the last 6 months
* BMI greater than or equal to 30.0 kg/m2
* Currently injecting in the thigh or abdomen
* HbA1c below 10%

Exclusion Criteria:

* Severe, uncontrolled hypertension
* Self-mixing insulin
* Unwillingness to monitor blood glucose
* Pregnancy, breast-feeding, intention to become pregnant, or inadequate contraceptive measures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2002-12; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 12 weeks of treatment

SECONDARY OUTCOMES:
Subject preference and handling
Frequency of hypoglycaemic episodes
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- United States (5):
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, San Antonio, Texas

REFERENCES:
- [Result] Schwartz S, Hassman D, Shelmet J, Sievers R, Weinstein R, Liang J, Lyness W. A multicenter, open-label, randomized, two-period crossover trial comparing glycemic control, satisfaction, and preference achieved with a 31 gauge x 6 mm needle versus a 29 gauge x 12.7 mm needle in obese patients with diabetes mellitus. Clin Ther. 2004 Oct;26(10):1663-78. doi: 10.1016/j.clinthera.2004.10.007. PMID 15598483
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com